CLINICAL TRIAL: NCT01138774
Title: Cellular and Molecular Effects of Lipoic Acid and Eicosapentaenoic Acid (EPA) on Adipose Tissue: Potential Application in Human Obesity
Brief Title: Effects of Lipoic Acid and Eicosapentaenoic Acid (EPA) in Human Obesity
Acronym: OBEPALIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBEPALIP
Record Dates: First submitted 2010-05-21; First posted 2010-06-07 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2012-02

CONDITIONS: Obesity; Body Fat; Insulin Resistance
Keywords: Obesity; Calorie restriction; Eicosapentaenoic acid (EPA); Lipoic acid; Weight loss; Insulin sensitivity; Lipid metabolism; Adipokines; Inflammation; Oxidative stress; Adipose tissue gene profile; Metabolomic profile
MeSH Terms: conditions — Obesity; Insulin Resistance; Weight Loss; Inflammation | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (Placebo Comparator): Dietary treatment with a calorie restriction of 30 % the subject's energy expenditure at baseline + placebos supplements
  Interventions: Dietary Supplement: Double blind dietary intervention with EPA and lipoic acid
- EPA group (Experimental): Dietary treatment with a calorie restriction of 30 % the subject's energy expenditure at baseline + EPA (1.3 g/day, 3 capsules of 433 mg/day) supplement (EPA Group).
  Interventions: Dietary Supplement: Double blind dietary intervention with EPA and lipoic acid
- Lipoic acid group (Experimental): Dietary treatment with a calorie restriction of 30 % the subject's energy expenditure at baseline + LA (300 mg/day, 3 capsules of 100 mg/day) supplement (LA Group)
  Interventions: Dietary Supplement: Double blind dietary intervention with EPA and lipoic acid
- EPA+LA group (Experimental): Dietary treatment with a calorie restriction of 30 % the subject's energy expenditure at baseline + EPA/LA (1.3 g /day and 300 mg/day respectively).
  Interventions: Dietary Supplement: Double blind dietary intervention with EPA and lipoic acid

INTERVENTIONS:
Dietary Supplement: Double blind dietary intervention with EPA and lipoic acid — Placebo-controlled dietary intervention during 10 weeks. All groups will have a dietary treatment with a calorie restriction of 30 % the subject's energy expenditure at baseline, supplemented with eicosapentaenoic acid (EPA) and/or lipoic acid (LA).

SUMMARY:
The aim of the study is to analyze the effects of Lipoic acid and/or EPA supplementation on weight loss, lipid profile, insulin resistance, oxidative and inflammation parameters, metabolomic profile as well as on adipose tissue gene profile in healthy overweight/obese subjects following an energy-restricted diet.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Ages between 20 and 45 years, and with regular menstrual cycles
* Body Mass Index (BMI) between 27.5 and 39.9 kg/m2
* Weight unchanged (± 3 kg) for the last 3 months
* All subjects should have an overall physical and psychological condition that the investigator believes is in accordance with the overall aim of the study.

Exclusion Criteria:

* Use of prescription medication
* To suffer from any chronic metabolic or obesity related disease, hepatic or renal systemic disease: Hypertension, dislipidemia, type 1 or 2 diabetes, thyroid function disorders, cirrhosis, fatty liver, etc.
* Food allergies or food intolerance expected to come up during the study
* Special diets (Atkins, vegetarian, etc.) prior three months the start of the study.
* Eating disorders
* Surgically treated obesity
* Pregnant or lactating women or planning to be pregnant in the next two months
* Alcohol or drug abuse (based on clinical parameters)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Weight Loss | Week 0 (baseline)
  Volunteers will attend the Nutritional Intervention unit (University of Navarra), where their weight will be measured to the nearest 0.1 kg.
Weight Loss | Week 2
  Volunteers will attend the Nutritional Intervention unit (University of Navarra), where their weight will be measured to the nearest 0.1 kg.
Weight Loss | Week 4
  Volunteers will attend the Nutritional Intervention unit (University of Navarra), where their weight will be measured to the nearest 0.1 kg.
Weight Loss | week 6
  Volunteers will attend the Nutritional Intervention unit (University of Navarra), where their weight will be measured to the nearest 0.1 kg.
Weight Loss | Week 8
  Volunteers will attend the Nutritional Intervention unit (University of Navarra), where their weight will be measured to the nearest 0.1 kg.
Weight Loss | Week 10 (end of treatment)
  Volunteers will attend the Nutritional Intervention unit (University of Navarra), where their weight will be measured to the nearest 0.1 kg.
Body composition and Anthropometric parameters | Week 0 (Baseline)
  Changes in body composition will be analyzed by Dual X-ray Absorptiometry (DXA) and by bioimpedance, and hip and waist circumferences will be measured.
Body composition and anthropometric parameters | Week 10 (end of treatment)
  Changes in body composition will be analyzed by Dual X-ray Absorptiometry (DXA) and by bioimpedance, and hip and waist circumferences will be measured.
Glucose metabolism parameters | Week 0 (baseline)
  Fasting serum glucose, Fasting serum insulin, Oral Glucose Tolerance Test, HOMA index
Glucose metabolism parameters | Week 10 (end of treatment)
  Fasting serum glucose, Fasting serum insulin, Oral Glucose Tolerance Test, HOMA index
Lipid metabolism biomarkers | Week 0 (baseline)
  Serum total-cholesterol, HDL-cholesterol, LDL-cholesterol, triacylglycerols, free fatty acids, ketone bodies.
Lipid metabolism biomarkers | Week 10 (end of treatment)
  Serum total-cholesterol, HDL-cholesterol, LDL-cholesterol, triacylglycerols, free fatty acids, ketone bodies.

SECONDARY OUTCOMES:
Blood Pressure and Cardiovascular Risk biomarkers | Baseline
  Blood pressure, PAI-1 and VEGF will be measured.
Blood Pressure and Cardiovascular Risk biomarkers | Week 10 (end of treatment)
  Blood pressure, PAI-1 and VEGF will be measured.
Energy expenditure | Baseline
  Energy expenditure will be estimated by indirect calorimetry, and T3, T4 and TSH levels will be analysed by ELISA kits
Energy expenditure | Week 10 (end of treatment)
  Energy expenditure will be estimated by indirect calorimetry, and T3, T4 and TSH levels will be analysed by ELISA kits
Satiety | Baseline
  Satiety will be estimated by using a VAS questionnaire
Satiety | Week 10 (end of treatment)
  Satiety will be estimated by using a VAS questionnaire
Serum inflammation biomarkers | Baseline
  TNF-alpha, IL-6, C-reactive protein, serum A-amiloid, Leptin, Adiponectin, Visfatin
Serum inflammation biomarkers | Week 10 (end of treatment)
  TNF-alpha, IL-6, C-reactive protein, serum A-amiloid, Leptin, Adiponectin, Visfatin
Serum oxidative stress biomarkers | Baseline
  Total and Reduced Glutathione, Glutathione Peroxidase, MDA, Superoxide Dismutase-2 (Mn-SOD).
Serum oxidative stress biomarkers | Week 10 (end of treatment)
  Total and Reduced Glutathione, Glutathione Peroxidase, MDA, Superoxide Dismutase-2 (Mn-SOD).
Adipose tissue gene profile and function analysis | Week 10 (end of treatment)
  A biopsy (2 g) of subcutaneous abdominal periumbilical area adipose tissue will be obtained. In order to identify clusters/pathways of genes regulated by the supplementation of EPA and LA, microarray gene profiling will be performed in adipose tissue from the 4 groups after the nutritional intervention. If possible primary explant culture of adipose tissue biopsies will be also carried out.
Metabolomic and lipidomic profile | Baseline
  Samples of plasma and 24-h urine will be analysed by Ultra Performance Liquid Chromatography-Mass Spectrometry (UPLC-MS), and Nuclear Magnetic Resonance (NMR), and Bidimensional Gas Chromatography-Mass Spectrometry (BC-MS).
Metabolomic and lipidomic profile | Week 10 (end of treatment)
  Samples of plasma and 24-h urine will be analysed by Ultra Performance Liquid Chromatography-Mass Spectrometry (UPLC-MS), and Nuclear Magnetic Resonance (NMR), and Bidimensional Gas Chromatography-Mass Spectrometry (BC-MS).

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Moreno-Aliaga, PhD, Principal Investigator — University of Navarra; Alfredo Martínez, PhD, Study Director — University of Navarra; Santiago Navas-Carretero, PhD, Study Chair — University of Navarra
Locations (1):
- Department of Nutrition, Food Science, Physiology and Toxicology. University of Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Prieto-Hontoria PL, Perez-Matute P, Fernandez-Galilea M, Barber A, Martinez JA, Moreno-Aliaga MJ. Lipoic acid prevents body weight gain induced by a high fat diet in rats: effects on intestinal sugar transport. J Physiol Biochem. 2009 Mar;65(1):43-50. doi: 10.1007/BF03165968. PMID 19588730
- [Background] Lorente-Cebrian S, Bustos M, Marti A, Martinez JA, Moreno-Aliaga MJ. Eicosapentaenoic acid up-regulates apelin secretion and gene expression in 3T3-L1 adipocytes. Mol Nutr Food Res. 2010 May;54 Suppl 1:S104-11. doi: 10.1002/mnfr.200900522. PMID 20352620
- [Background] Lorente-Cebrian S, Bustos M, Marti A, Martinez JA, Moreno-Aliaga MJ. Eicosapentaenoic acid stimulates AMP-activated protein kinase and increases visfatin secretion in cultured murine adipocytes. Clin Sci (Lond). 2009 Aug 14;117(6):243-9. doi: 10.1042/CS20090020. PMID 19296827
- [Background] Perez-Echarri N, Perez-Matute P, Marcos-Gomez B, Marti A, Martinez JA, Moreno-Aliaga MJ. Down-regulation in muscle and liver lipogenic genes: EPA ethyl ester treatment in lean and overweight (high-fat-fed) rats. J Nutr Biochem. 2009 Sep;20(9):705-14. doi: 10.1016/j.jnutbio.2008.06.013. Epub 2008 Sep 30. PMID 18829285
- [Background] Perez-Echarri N, Perez-Matute P, Marcos-Gomez B, Baena MJ, Marti A, Martinez JA, Moreno-Aliaga MJ. Differential inflammatory status in rats susceptible or resistant to diet-induced obesity: effects of EPA ethyl ester treatment. Eur J Nutr. 2008 Oct;47(7):380-6. doi: 10.1007/s00394-008-0738-3. Epub 2008 Sep 18. PMID 18807107
- [Background] Perez-Echarri N, Perez-Matute P, Marcos-Gomez B, Martinez JA, Moreno-Aliaga MJ. Effects of eicosapentaenoic acid ethyl ester on visfatin and apelin in lean and overweight (cafeteria diet-fed) rats. Br J Nutr. 2009 Apr;101(7):1059-67. doi: 10.1017/S0007114508048307. Epub 2008 Aug 28. PMID 18755047
- [Background] Perez-Matute P, Perez-Echarri N, Martinez JA, Marti A, Moreno-Aliaga MJ. Eicosapentaenoic acid actions on adiposity and insulin resistance in control and high-fat-fed rats: role of apoptosis, adiponectin and tumour necrosis factor-alpha. Br J Nutr. 2007 Feb;97(2):389-98. doi: 10.1017/S0007114507207627. PMID 17298710
- [Background] Marrades MP, Martinez JA, Moreno-Aliaga MJ. Differences in short-term metabolic responses to a lipid load in lean (resistant) vs obese (susceptible) young male subjects with habitual high-fat consumption. Eur J Clin Nutr. 2007 Feb;61(2):166-74. doi: 10.1038/sj.ejcn.1602500. Epub 2006 Aug 9. PMID 16900083
- [Background] Marrades MP, Milagro FI, Martinez JA, Moreno-Aliaga MJ. Differential expression of aquaporin 7 in adipose tissue of lean and obese high fat consumers. Biochem Biophys Res Commun. 2006 Jan 20;339(3):785-9. doi: 10.1016/j.bbrc.2005.11.080. Epub 2005 Nov 22. PMID 16325777
- [Background] Ramel A, Martinez A, Kiely M, Morais G, Bandarra NM, Thorsdottir I. Beneficial effects of long-chain n-3 fatty acids included in an energy-restricted diet on insulin resistance in overweight and obese European young adults. Diabetologia. 2008 Jul;51(7):1261-8. doi: 10.1007/s00125-008-1035-7. Epub 2008 May 20. PMID 18491071
- [Background] Parra D, Ramel A, Bandarra N, Kiely M, Martinez JA, Thorsdottir I. A diet rich in long chain omega-3 fatty acids modulates satiety in overweight and obese volunteers during weight loss. Appetite. 2008 Nov;51(3):676-80. doi: 10.1016/j.appet.2008.06.003. Epub 2008 Jun 14. PMID 18602429
- [Background] Ramel A, Martinez JA, Kiely M, Bandarra NM, Thorsdottir I. Moderate consumption of fatty fish reduces diastolic blood pressure in overweight and obese European young adults during energy restriction. Nutrition. 2010 Feb;26(2):168-74. doi: 10.1016/j.nut.2009.04.002. Epub 2009 May 31. PMID 19487105
- [Background] Navas-Carretero S, Perez-Granados AM, Schoppen S, Vaquero MP. An oily fish diet increases insulin sensitivity compared to a red meat diet in young iron-deficient women. Br J Nutr. 2009 Aug;102(4):546-53. doi: 10.1017/S0007114509220794. Epub 2009 Feb 12. PMID 19210857
- [Derived] Romo-Hualde A, Huerta AE, Gonzalez-Navarro CJ, Ramos-Lopez O, Moreno-Aliaga MJ, Martinez JA. Untargeted metabolomic on urine samples after alpha-lipoic acid and/or eicosapentaenoic acid supplementation in healthy overweight/obese women. Lipids Health Dis. 2018 May 9;17(1):103. doi: 10.1186/s12944-018-0750-4. PMID 29743087
- [Derived] Huerta AE, Prieto-Hontoria PL, Sainz N, Martinez JA, Moreno-Aliaga MJ. Supplementation with alpha-Lipoic Acid Alone or in Combination with Eicosapentaenoic Acid Modulates the Inflammatory Status of Healthy Overweight or Obese Women Consuming an Energy-Restricted Diet. J Nutr. 2015 Apr 1;146(4):889S-896S. doi: 10.3945/jn.115.224105. PMID 26962183
- See also: European Master´s Degree in Feeding, Nutrition and Metabolism — http://www.unav.es/master/nutricion-metabolismo/